CLINICAL TRIAL: NCT02510495
Title: Effect of Different Endoscopic Papillary Balloon Dilation Duration Time on Complications of Common Bile Duct Stone Patient
Brief Title: Effect of Endoscopic Papillary Balloon Dilation on ERCP Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Xun Li, Professor of surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ERCP Balloon Dilation
Record Dates: First submitted 2015-07-20; First posted 2015-07-29 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Complications
Keywords: Sphincterotomy; Dilatation; Common bile duct; Pancreatitis
MeSH Terms: conditions — Dilatation, Pathologic; Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 0" group (No Intervention): After a small sphincterotomy was performed, a controlled radial expansion (CRE) balloon (diameter 8, 9, 10, 11, 12, 13.5, 15; Boston Scientific) was chosen according to the diameter of bile duct. It was placed across the papilla orifice and then gradually filled with diluted contrast in 15 seconds. When the waist disappeared, the balloon was deflated immediately. The stones were then retrieved by a basket or retrieval balloon. Mechanical lithotripsy was used if necessary.
- 30" group (Experimental): After a small sphincterotomy was performed, a controlled radial expansion (CRE) balloon (diameter 8, 9, 10, 11, 12, 13.5, 15; Boston Scientific) was chosen according to the diameter of bile duct. It was placed across the papilla orifice and then gradually filled with diluted contrast in 15 seconds. When the waist disappeared, the balloon was inflated till 30 seconds prior deflated. The stones were then retrieved by a basket or retrieval balloon. Mechanical lithotripsy was used if necessary.
  Interventions: Procedure: 30" group
- 60" group (Experimental): After a small sphincterotomy was performed, a controlled radial expansion (CRE) balloon (diameter 8, 9, 10, 11, 12, 13.5, 15; Boston Scientific) was chosen according to the diameter of bile duct. It was placed across the papilla orifice and then gradually filled with diluted contrast in 15 seconds. When the waist disappeared, the balloon was inflated till 60 seconds prior deflated. The stones were then retrieved by a basket or retrieval balloon. Mechanical lithotripsy was used if necessary.
  Interventions: Procedure: 60" group
- 180" group (Experimental): After a small sphincterotomy was performed, a controlled radial expansion (CRE) balloon (diameter 8, 9, 10, 11, 12, 13.5, 15; Boston Scientific) was chosen according to the diameter of bile duct. It was placed across the papilla orifice and then gradually filled with diluted contrast in 15 seconds. When the waist disappeared, the balloon was inflated till 180 seconds prior deflated. The stones were then retrieved by a basket or retrieval balloon. Mechanical lithotripsy was used if necessary.
  Interventions: Procedure: 180" group
- 300" group (Experimental): After a small sphincterotomy was performed, a controlled radial expansion (CRE) balloon (diameter 8, 9, 10, 11, 12, 13.5, 15; Boston Scientific) was chosen according to the diameter of bile duct. It was placed across the papilla orifice and then gradually filled with diluted contrast in 15 seconds. When the waist disappeared, the balloon was inflated till 300 seconds prior deflated. The stones were then retrieved by a basket or retrieval balloon. Mechanical lithotripsy was used if necessary.
  Interventions: Procedure: 300" group

INTERVENTIONS:
Procedure: 30" group — A small sphincterotomy (EST) was performed prior to the EPBD, the length of a small sphincterotomy was considered as no larger than the range which from the orifice to the top one-third of the papilla. a CRE balloon (diameter 8, 9, 10, 11, 12, 13.5, 15; Boston Scientific) was chosen according to the diameter of bile duct. It was placed across the papilla orifice and then gradually filled with diluted contrast in 15 seconds. When the waist disappeared, the balloon was inflated till 30 seconds prior deflated. The stones were then retrieved by a basket or retrieval balloon. Mechanical lithotripsy was used if necessary.
  Arms: 30" group
Procedure: 60" group — A small sphincterotomy (EST) was performed prior to the EPBD, the length of a small sphincterotomy was considered as no larger than the range which from the orifice to the top one-third of the papilla. a CRE balloon (diameter 8, 9, 10, 11, 12, 13.5, 15; Boston Scientific) was chosen according to the diameter of bile duct. It was placed across the papilla orifice and then gradually filled with diluted contrast in 15 seconds. When the waist disappeared, the balloon was inflated till 60 seconds prior deflated. The stones were then retrieved by a basket or retrieval balloon. Mechanical lithotripsy was used if necessary.
  Arms: 60" group
Procedure: 180" group — A small sphincterotomy (EST) was performed prior to the EPBD, the length of a small sphincterotomy was considered as no larger than the range which from the orifice to the top one-third of the papilla. a CRE balloon (diameter 8, 9, 10, 11, 12, 13.5, 15; Boston Scientific) was chosen according to the diameter of bile duct. It was placed across the papilla orifice and then gradually filled with diluted contrast in 15 seconds. When the waist disappeared, the balloon was inflated till 180 seconds prior deflated. The stones were then retrieved by a basket or retrieval balloon. Mechanical lithotripsy was used if necessary.
  Arms: 180" group
Procedure: 300" group — A small sphincterotomy (EST) was performed prior to the EPBD, the length of a small sphincterotomy was considered as no larger than the range which from the orifice to the top one-third of the papilla. a CRE balloon (diameter 8, 9, 10, 11, 12, 13.5, 15; Boston Scientific) was chosen according to the diameter of bile duct. It was placed across the papilla orifice and then gradually filled with diluted contrast in 15 seconds. When the waist disappeared, the balloon was inflated till 300 seconds prior deflated. The stones were then retrieved by a basket or retrieval balloon. Mechanical lithotripsy was used if necessary.
  Arms: 300" group

SUMMARY:
The purpose of this study is to determine how different endoscopic papillary balloon dilatation (EPBD) duration time affects the complications after endoscopic retrograde cholangiopancreatography (ERCP) in the treatment of common bile duct stones.

DETAILED DESCRIPTION:
Common bile duct (CBD) stone is a common disease with high morbidity. Half century ago, surgery with bile duct exploration and T-tube drainage was the only radical treatment for the stones until a revolutionary technique was reported in 1970, which possible to remove stone by means of endoscopic sphincterotomy (EST) during endoscopic retrograde cholangiopancreatography (ERCP). Since then, EST became a very promising measure for both patients and doctors to meet the purpose of minimally invasive treatment. However, EST remains an advanced technique which requires high skills of the endoscopist. As far as patients who have anatomical biliary abnormalities, such as papillary diverticulum, are more likely to end up with severe complications such as bleeding and perforation during EST procedure. On the other hand, EST may also lead to permanent dysfunction of the Oddi's sphincter. It is currently reported that a growing number of young patients, even some children are managed with EST which is still debated due to the existence of some long-term complications.

Endoscopic papillary balloon dilatation (EPBD) is an alternative technique developed to achieve the same purpose as EST but preserving Oddi's sphincter' function partially, and more than that, EPBD is easy to grasp for endoscopist. By using a columnar balloon, Oddi's sphincter can be expanded without direct transection, and the temporary relaxation of Oddi's sphincter makes it possible to remove the stones and the rest of the procedures as well. Removing common bile duct stone by EPBD was firstly reported in 1982 and proved to be safe and efficient. However, clinical observations have been found that simple EPBD has a higher incidence of developing acute pancreatitis after ERCP, especially in patients with intact papilla. The speculated reason for high post-ERCP pancreatitis (PEP) rate might be pancreatic duct orifice edema resulted from inadequate destroy of Oddi's sphincter during a balloon dilatation, leading the pancreatic duct obstructed and high ductal pressure afterward. Retrospective study has indicated the PEP rate of post-EPBD by 10% which was considered slightly higher than ordinary EST before a new modified method has been introduced by a small EST prior to EPBD. Currently small EST plus EPBD has been increasingly used in clinical and proven to be an effective treatment for improving the success rate of the common bile duct stone removal, preserving Oddi's sphincter function and lowering long-term complications.

Dedicate practitioners conducted many kinds of studies about reducing post-ERCP complications, and nowadays, some of them focus on the dilation time of EPBD which would be suspected as the key point of the issues. Nonetheless, more institutes are willing to join in EPBD research as the universal concerns for post-ERCP complications increases, no common agreements achieved at present.

From some prospected data, we might see confused results. Slowly inject balloon with a contrast agent and keep dilating for 1-2 minutes, until 15 seconds after the image of papilla and balloon waist disappeared is able to get the same stone removal rate as regular procedure does, and a slower balloon filling performance is helpful to protect the Oddi's sphincter function and reduce post-ERCP complications. However, other studies conclude there are no difference no matter in stone removal rate or post-ERCP pancreatitis instead of blood amylase, in which arms are 20 seconds compared 60 seconds and 30 seconds compared 60 seconds. Interestingly, there is another inspiring randomized controlled trial (RCT) study which prolong the dilation time up to 5 minutes. The author figured that PEP rate of five minutes group is smaller than that of the 1-minute group as well as stone removal.

Few studies concerning the optimal duration time of EPBD which is very important to patients' safety and maximum utilization of the easier handled EPBD procedure compared to EST. Therefore this large volume multicenter prospective randomize control study targets on how different EPBD duration management affect the complications after ERCP which attempts to discover a promising method for safe therapy in common bile duct stones.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* CBD stone patients, stone diameter≤1.5cm, CBD diameter≤2cm

Exclusion Criteria:

* Unwillingness or inability to consent for the study
* Coagulation dysfunction (INR> 1.3) and low peripheral blood platelet count (<50×109 / L) or using anti-coagulation drugs
* Previous EST or EPBD
* Prior surgery of Bismuth Ⅱ and Roux-en-Y
* Benign or malignant CBD stricture
* Preoperative coexistent diseases: acute pancreatitis, GI tract hemorrhage, severe liver disease, primary sclerosing cholangitis (PSC), septic shock
* Combined with Mirizzi syndrome and intrahepatic bile duct stones
* Malignant disease
* Biliary-duodenal fistula confirmed during ERCP
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1920 (Actual)
Dates: Start 2016-02; Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Post-ERCP pancreatitis | Within 7 days after ERCP
  Upper abdominal pain with serum amylase elevation no less than 462 U/L after the procedure

SECONDARY OUTCOMES:
Hemorrhage | Within 7 days after ERCP
  Maintained positive fecal occult blood test appears
Perforation | Within 7 days after ERCP
  CT scan shows retroperitoneal space fluid or gas
Acute cholangitis | Within 7 days after ERCP
  Intermittent chills and fever after ERCP
Pain | Within 7 days after ERCP
  Upper abdominal pain after ERCP measured by Numerical Rating Scale
Operation time | Up to 2 hours
  From successful biliary intubation to end of operation
Average hospital stay | Up to 30 days
  Length of stay in hospital
Stone clearance rate | Up to 2 hours
  The proportion of patients with all stones removed
Success rate of stone extraction in the initial attempt | Up to 2 hours
  The proportion of patients with all stones removed in first attempt after EPBD
Rate of mechanical lithotripsy | Up to 2 hours
  The proportion of patients whose stones need mechanical lithotripsy before removed
X-ray exposure time | Up to 2 hours
  The total radiography time during ERCP
Pancreatic duct insertion times | Up to 2 hours
  Times of any accessories goes into the pancreatic duct, no matter how depth

CONTACTS AND LOCATIONS:
Overall Officials: Xun Li, M.D., Ph.D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (15):
- China (15):
  - Third Military Medical University, Chongqing, Chongqing Municipality
  - The first hospital of Lanzhou university, Lanzhou, Gansu
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Union hospital,Tongji medical collage,Huazhong University of science and technology, Wuhan, Hubei
  - Second Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The first affiliated hospital of Xi 'an jiaotong university, Xi'an, Shaanxi
  - Shandong jiaotong Hospital, Jinan, Shandong
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Taiyuan Iron and Steel Corporation Hospital, Taiyuan, Shanxi
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Tianjin Nankai Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meine GC, Baron TH. Endoscopic papillary large-balloon dilation combined with endoscopic biliary sphincterotomy for the removal of bile duct stones (with video). Gastrointest Endosc. 2011 Nov;74(5):1119-26; quiz 1115.e1-5. doi: 10.1016/j.gie.2011.06.042. Epub 2011 Sep 23. No abstract available. PMID 21944309
- [Background] Tsujino T, Kawabe T, Komatsu Y, Yoshida H, Isayama H, Sasaki T, Kogure H, Togawa O, Arizumi T, Matsubara S, Ito Y, Nakai Y, Yamamoto N, Sasahira N, Hirano K, Toda N, Tada M, Omata M. Endoscopic papillary balloon dilation for bile duct stone: immediate and long-term outcomes in 1000 patients. Clin Gastroenterol Hepatol. 2007 Jan;5(1):130-7. doi: 10.1016/j.cgh.2006.10.013. PMID 17234559
- [Background] Bang BW, Jeong S, Lee DH, Lee JI, Lee JW, Kwon KS, Kim HG, Shin YW, Kim YS. The ballooning time in endoscopic papillary balloon dilation for the treatment of bile duct stones. Korean J Intern Med. 2010 Sep;25(3):239-45. doi: 10.3904/kjim.2010.25.3.239. Epub 2010 Aug 31. PMID 20830219
- [Background] Ozaslan E. Comment to "Sixty- versus thirty-seconds papillary balloon dilation after sphincterotomy for the treatment of large bile duct stones: a randomized controlled trial". Dig Liver Dis. 2013 Aug;45(8):700. doi: 10.1016/j.dld.2013.02.004. Epub 2013 Mar 13. No abstract available. PMID 23490342
- [Background] Liao WC, Lee CT, Chang CY, Leung JW, Chen JH, Tsai MC, Lin JT, Wu MS, Wang HP. Randomized trial of 1-minute versus 5-minute endoscopic balloon dilation for extraction of bile duct stones. Gastrointest Endosc. 2010 Dec;72(6):1154-62. doi: 10.1016/j.gie.2010.07.009. Epub 2010 Sep 25. PMID 20869710
- [Derived] Meng W, Leung JW, Zhang K, Zhou W, Wang Z, Zhang L, Sun H, Xue P, Liu W, Wang Q, Zhang J, Wang X, Wang M, Shao Y, Cai K, Hou S, Li Q, Zhang L, Zhu K, Yue P, Wang H, Zhang M, Sun X, Yang Z, Tao J, Wen Z, Wang Q, Chen B, Shao Q, Zhao M, Zhang R, Jiang T, Liu K, Zhang L, Chen K, Zhu X, Zhang H, Miao L, Wang Z, Li J, Yan X, Wang F, Zhang L, Suzuki A, Tanaka K, Nur U, Weiderpass E, Li X. Optimal dilation time for combined small endoscopic sphincterotomy and balloon dilation for common bile duct stones: a multicentre, single-blinded, randomised controlled trial. Lancet Gastroenterol Hepatol. 2019 Jun;4(6):425-434. doi: 10.1016/S2468-1253(19)30075-5. Epub 2019 Apr 16. PMID 31003961